CLINICAL TRIAL: NCT04968587
Title: Comparison of Regional Citrate Anticoagulation (RCA) and Regional Anticoagulation by Citrate-Free Decalcification in Renal (RACD) Replacement Therapy Using Sustained Low-Efficiency Dialysis
Brief Title: Comparison of RCA and RACD in Extra-renal Purification by SLED
Acronym: ARDC-SLED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Sud Ile-de-France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-A0122-37
Record Dates: First submitted 2021-06-08; First posted 2021-07-20 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Hybrid Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: RACD - RCA (Other): First period of treatment with Regional Anticoagulation by Citrate-Free Decalcification SLED and second period of treatment with Regional Citrate Anticoagulation SLED
  Interventions: Procedure: Sustained Low-Efficiency Dialysis
- Group 2 : RCA - RACD (Other): First period of treatment with Regional Citrate Anticoagulation SLED and second period of treatment with Regional Anticoagulation by Citrate-Free Decalcification SLED
  Interventions: Procedure: Sustained Low-Efficiency Dialysis

INTERVENTIONS:
Procedure: Sustained Low-Efficiency Dialysis — All patient requiring Renal replacement Therapy in the intensive care unit will be randomized in open order (cross-over) with either Regional anticoagulation with Citrate or Regional anticoagulation by Decalcification without Citrate
  Other Names: intermittent haemodialysis equipment with lower blood flow and dialysate flow combined with prolonged sessions

SUMMARY:
One of the main RRT issues is anticoagulation of the ECC, because blood contact with biomaterials causes bio-incompatibility reactions, including activation of the coagulation cascade. Based on Regional Citrate Anticoagulation (RCA) protocols, an ionized calcium (Ca-ion) concentration around 0.25 to 0.35mmol / L prevents fibrino formation and allows anticoagulation for the ECC. During RCA, metabolic side effects may occur due to systemic flow of citrate. Our postulate is that reduction of ionized calcemia related to the use of a calcium-free dialysate and haemofilter performance makes it possible to avoid citrate infusion. Our study aim to compare intermittent RRT using 4% Citrate infusion and without Citrate.

DETAILED DESCRIPTION:
Background: Renal Replacement Therapy (RRT), requires anticoagulation of the extracorporal circuit (ECC) using heparin, citrate or repeated rinsing. Difficulties of implementation or exposition to complications (thrombosis, hemorrhage or electrolyte disorder) are frequent.

Purpose: Regional anticoagulation of the ECC based on ionized calcemia reduction, as using citrate, but induced by the use of a calcium-free dialysate associated with the performance of the hemofilter could reduce these risks and the cost of intermittent RRT. This study aims to compare the efficiency of a regional anticoagulation technique based on the reduction of Ionized Calcium in the extracorporal circuit, without the use of Citrate and with Citrate during intermittent RRT.

Abstract: One of the main RRT issue is anticoagulation of the ECC, because blood contact with biomaterials causes bio-incompatibility reactions, including activation of the coagulation cascade. Based on Regional Citrate anticoagulation (RCA) protocols, an ionized calcium (Ca-ion) concentration around 0.25 to 0.35mmol/L prevents fibrino formation and allows anticoagulation for the ECC. During RCA, metabolic side effects may occur due to systemic passage of citrate. Our postulate is that reduction of ionized calcemia related to the use of a calcium-free dialysate and haemofilter performance makes it possible to avoid citrate infusion. Our study aims at comparing intermittent RRT using 4% Citrate infusion and without Citrate.

ELIGIBILITY:
Inclusion Criteria:

* All patient requiring Renal replacement Therapy

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Hypercalcemia ≥ 3 mmol/L.
* Major under guardianship
* Major deprived of freedom
* Impossible to obtain free and informed consent
* Presence of hemostasis or coagulation disorders:
* Thrombocytopenia < 30 G/L.
* Curative anticoagulation.
* Severe liver disease with Prothrombin rate <30%.
* Coagulation factor deficit.
* Not registered to a social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the plasma urea | up to 8 hours
  We will compare plasma urea clearance after reaching the prescribed session time without irreversible coagulation of the extracorporeal circuit, with both methods tested in the study.

SECONDARY OUTCOMES:
Measurement of the concentration of Ca²+i in post-filter | 30 minutes, 1 hour; 4 hours and 8 hours
  Measurement at different timepoints after the beginning of the concentration of Ca²+i in post-filter during each RRT session.
Measurement of the concentration of Ca²+i (patient) | 30minutes, 1 hour; 4 hours and 8 hours
  Measurement at different timepoints after the beginning of the concentration of Ca²+i (patient) during each RRT session.
Measurement of the concentration of Mg2+ | 8 hours
  Measurement of the concentration of Mg2+ at the end of each RRT session.
Measurement of heart rate during each RRT session. | Hour 0; 30 minutes; 60 minutes; 90 minutes; 120 minutes; 150 minutes; 180 minutes; 210 minutes; 240 minutes; 270 minutes; 300 minutes; 330 minutes; 360 minutes; 390 minutes; 420 minutes; 450 minutes; 480 minutes
  Measurement heart rate during each RRT session.
Measurement of blood pressure | Hour 0; 30 minutes; 60 minutes; 90 minutes; 120 minutes; 150 minutes; 180 minutes; 210 minutes; 240 minutes; 270 minutes; 300 minutes; 330 minutes; 360 minutes; 390 minutes; 420 minutes; 450 minutes; 480 minutes
  Measurement of blood pressure during each RRT session.
Number of circuit losses during each RRT session, | Hour 0; 480 minutes
  Number of circuit losses during each RRT sessions,
Number of catheter thrombosis during each RRT session | Hour 0; 480 minutes
  Number of catheter thrombosis during each RRT session

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Sud Ile-de-France, Melun, France

IPD SHARING:
Plan to Share IPD: No